CLINICAL TRIAL: NCT01660659
Title: Use of Biomass Briquettes: Its Effect on Indoor Air Pollution and on Pneumococcal Nasopharyngeal Carriage. A Randomized Clinical Trial
Brief Title: Indoor Air Pollution (IAP) Carriage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SCC 1284
Record Dates: First submitted 2012-05-18; First posted 2012-08-09 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Pneumococcal Carriage; Particulate Matter
Keywords: Indoor air pollution; pneumococcal carriage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cooking with Biomass Briquettes and Rocket Stove (Experimental): cooking with Biomass Briquettes and Rocket Stove
  Interventions: Device: Biomass Briquettes and Rocket stove
- standard cooking (No Intervention): standard way of cooking

INTERVENTIONS:
Device: Biomass Briquettes and Rocket stove — Biomass briquettes are made from dried peanut shells. Rocket stoves were designed to efficiently burn the briquettes
  Arms: cooking with Biomass Briquettes and Rocket Stove

SUMMARY:
Personal exposure to Indoor Air Pollution (IAP) is a known risk factor of severe pneumonia, which is the number one killer of children under five in developing countries. The main source of IAP in developing countries is cooking fires, with an estimated 3 billion people still reliant on biomass stoves for their daily cooking. This study will test the effectiveness of an intervention aimed to reduce IAP, as well as help to quantify the relationship between exposure (IAP) and infection (pneumococcal carriage).

In Phase I (adjunct pilot study L2010.99), 3 fuels and 5 stoves were tested to measure harmful pollutant emissions. The preliminary results showed that the largest difference was found in the fuels (briquettes cleaner than wood), with a smaller difference found between a couple of the improved stoves and the traditional 3-stone. Re-testing of selected stove/fuel combinations to confirm findings has just been completed. Phase II (this proposal) will test the biomass briquettes in a randomized clinical trial to measure actual IAP reductions in households. A proof of concept pneumococcal survey will also be conducted as a secondary study to see whether reduced exposure to IAP affects pneumococcal carriage in babies and mothers

DETAILED DESCRIPTION:
Acute respiratory infections (ARI), specifically Severe Pneumonia, are the leading cause of death in children under 5 years of age. Of the nearly 10 million children under 5 who die each year, 1.9 million die from ARI, almost all of which occur in developing countries [1, 2]. Over the years, various studies have identified many risk factors associated with ARI, including malnutrition, zinc deficiency, indoor air pollution (IAP) from solid fuels and tobacco. Proven efficacious interventions have been developed and studied to address risk factors related to nutrition and zinc deficiency but still little is known about IAP and proven effective interventions. Furthermore, little is known about the quantifiable relationship between IAP exposure and disease, specifically ARI.

IAP from cooking with biomass is one of the top ten global health risks [3]. 1.6 million people are estimated to die every year from IAP exposure, of which half of them are children under 5 years of age [4]. In developing countries, IAP is estimated to account for 3.7% of the total burden of disease, making it the fourth most serious health risk factor after malnutrition, STDs, and inadequate water and sanitation [5]. A recent meta-analysis found that children under 5 years old living in households using biomass fuels had a 78% greater chance of contracting pneumonia than did children in households with cleaner-burning fuels [6]. In Africa, 94% of the rural population and 73% of the urban population use solid fuels as their primary source of energy [7]. Not only does IAP disproportionally affect the poor, but it also affects women and children who spend more time near the cooking fires and are therefore are most exposed.

Because of the difficulty in measuring exposure, most observational studies use proxy measures. These proxies include the type of fuel used, amount of time spent near the cooking fires, or whether the child is carried on the mother's back during cooking. But because variations in personal exposure in most countries depend on a variety of factors (e.g. fuel, stove, housing, behavioral), proxy indicators are an insufficient method to effectively capture variations in exposure [8]. This affects the understanding and knowledge of the potential health gains that might result from reducing exposure by varying amounts. Determining this exposure-disease relationship is crucial to understanding the possible impacts that interventions may have on improving health [9]. Unfortunately, the amount of research being done on pollutant exposure from IAP is negligible compared to the huge disease burden associated with this exposure [10]. A lot more research needs to be conducted to help the lives of the 3 billion affected from these harmful pollutants.

Interventional Research Interventional research has focused on developing more efficient biomass stoves as an approach to reduce IAP, yet few studies have looked into alternative biomass fuels. Though improved stoves have shown to reduce pollutant emissions in controlled settings, it remains difficult to measure the true effectiveness of this intervention, i.e. whether these stoves are actually reducing pollutants in local kitchens. The Water Boiling Test (WBT) and Controlled Cooking Tests (CCT), both of which are conducted in controlled environments, are based on the assumption that performing a simple cooking task produces estimates that can be used when evaluating technology for developing populations [11]. However, because of the numerous behavioral and outside variables that can alter the efficiency of a stove, these tests do not illustrate the true picture of how the technology will perform among the population [12]. The Kitchen Performance Test (KPT) has been designed to measure the effectiveness though because of its difficulties in implementation, it is often not used to measure stove performance. Furthermore, there have been varying results in the field effectiveness of reducing IAP with improved stoves [9]. Given the wide variability in stoves and settings, it remains difficult to know what levels of IAP exposure reductions can be expected.

Because of the uncertainties and challenges of reducing IAP with improved stoves, other interventions to reduce pollutant levels need to be explored, such as the use of alternative biomass fuel in lieu of wood. A study in 2003 in rural Kenya looked at modelling potential reductions on disease following interventions including fuel, stove type and cooking location. This study showed that the largest reduction was from switching fuels and not stoves [3]. There are a handful of studies throughout developing countries that are currently looking at using crop waste as an alternative fuel. But because crop waste varies greatly with locality, separate testing needs be done on these different crop wastes and their transformation into cooking fuel. In The Gambia and most of West and Central Africa, groundnuts are a major cash crop and their shells are available in abundance. Recently, two separate factories have been established in The Gambia to process these dried groundnut shells into biomass briquettes, which will then be used as cooking fuel. During Phase I of this study, the investigators have tested (and are currently retesting) the two available biomass briquettes made from groundnut shells. Both the WBT and CCT are being conducted to evaluate the performance of these fuels (in comparison to wood and charcoal) when used with different stoves, as well as IAP emissions. These tests were conducted in accordance with the protocol developed for the Shell Foundation and Household Energy Health Program [13, 14]. The investigators also concurrently measured PM2.5 concentrations two ways: continuous PM2.5 concentrations using light-scattering, TSI 8520 DustTrak monitors and integrated PM2.5 concentrations using gravimetric Casella pumps, cyclones, and Teflon filters. CO concentrations were also measured alongside the CCT using Drager CO 50/a-D Diffusion Tubes. The Investigators preliminary analysis shows that the briquettes do burn much cleaner than wood when used with each of the tested stoves. The investigators are currently retesting the briquettes with the different stoves to assure the investigators have the cleanest stove/fuel combination for Phase II.

For Phase II (this proposal), the investigators will test the effectiveness of the biomass briquettes in the communities. It is possible the investigators will also use an improved stove with the briquettes, though this decision will not be made until the final analysis is complete in December/January. However, based on the preliminary analysis, the investigators are leaning more towards briquettes with the traditional 3-stone. For simplicity sake, briquettes are mentioned as the intervention throughout this document. Though RCTs usually measure the efficacy of an intervention, this study is slightly different in that the efficiency and efficacy have already been conducted in Phase I. This study will enable the investigators to evaluate the true reduction of IAP emissions in the study population, as well as the cost effectiveness of using briquettes compared to wood or charcoal. From the preliminary research, the investigators found that the briquettes performed very similarly to wood, and therefore do not anticipate difficulties in adopting the use of briquettes.

Using pneumococcal carriage as a proxy measure for a health outcome Pneumonia accounts for ~30% of deaths of children under the age of 5 in developing countries, most resulting from Streptococcus pneumoniae (pneumococcus). Pneumococci generally colonizes the nasopharynx within the first months of life, with carriage rates in children in developing countries 2-3 times higher than those found in children from developed countries[15, 16]. In one study in The Gambia, it was found that pneumococcal carriage was greater than 80% during the third month of life [17]. In another study in Bangladesh, it was found that 50% of the children had been colonized by pneumococci at least once by the age of 8 weeks [18]. Though pneumococcal carriage is present in many healthy people, it is an identifiable risk for disease, predominantly affecting the young in developing countries.

Nasopharyngeal colonization is a necessary phase before infection with S pneumoniae can occur [19]. Therefore, preventing colonization from ever happening can be an important measure to preventing S pneumoniae. As IAP exposure is one major risk factor to developing ARI, understanding how IAP exposure can affect the risk of infection for pneumococcal carriers can help us better understand the quantitative relationship between IAP exposure and disease (severe pneumonia). There have been previous studies looking at the impact tobacco smoke has on carriage, but to date, there has yet to be any research done looking at carriage and IAP exposure. This study may be instrumental in helping understand this complex exposure-disease relationship. This component of the study is a Proof-of-Concept study, and is therefore designed to illustrate the potential relationship between IAP exposure and ARI. If using pneumococcal carriage as a proxy does show to be an effective tool in helping to quantify the this relationship, it has the potential to lay the foundation for further research looking at IAP and its affect on pneumococcal carriage.

ELIGIBILITY:
Inclusion Criteria:

* Child between 2 to 8 months of age at start of the study (1st pneumococcal swab)
* residing within the catchment area
* the mother relies only on wood and the 3-stone stove for all her cooking
* the mother will cook in an indoor kitchen only (not outside; 4 walls with a roof)
* written informed consent

Exclusion Criteria:

* will be traveling from their home during the following 6 months
* already involved in another study

Ages: 2 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
IAP Carriage Study | 12 months
  1. Integrated PM2.5 concentrations (48 hour measurements in each kitchen) Integrated PM2.5 concentrations will be measured using gravimetric Casella and SKC pumps, cyclones, and Teflon filters. The pumps will run one minute on, 5 minutes off, for 48 continuous hours in each of the participating cookhouses. These integrated measurements will allow us to compare the emissions from briquettes and firewood.
  The measurements will take place at a random time during the 16 week invention period

SECONDARY OUTCOMES:
IAP Carriage Study | 12 months
  To measure the prevalence of pneumococcal carriage in both study arms. These surveys will occur at the start of the study (before the intervention) to capture the baseline measurement, and at the end of the study (after the 16 weeks of intervention), to see whether reduced exposure to PMs affects pneumococcal carriage in the mothers and babies

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Litchfield, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Medical Research Council Unit, Fajara, The Gambia